CLINICAL TRIAL: NCT00172939
Title: Molecular Mechanisms of Helium-Neon Laser on Melanocyte Regeneration in Skin Equivalent Vitiligo Model
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9461700332
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-03

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

INTERVENTIONS:
Procedure: foreskin from healthy adults

SUMMARY:
This current three-year proposal aims to clarify the mechanisms of melanocyte destruction and regeneration in vitiligo lesions using both traditional cell culture and skin equivalent model (organotypic culture).

DETAILED DESCRIPTION:
Melanocytes (MCs) are melanin-producing cells of the skin that are derived from neural crest cells. Vitiligo vulgaris is a common depigmentation disorder resulting from destruction of functional MCs in the affected skin. Although this disorder affects all races and occurs in approximately 1% of the world population, its pathogenesis remains obscure. Recovery from vitiligo is initiated by the activation, proliferation, and migration of melanoblasts (MBs) to the epidermis. The subsequent maturation of MBs leads to production of melanosomes that will be transferred to the juxtaposed keratinocytes. The beam of a low-energy laser produces a temperature elevation of less than 0.5 ℃. Therefore, light-mediated reaction by such laser irradiation is referred to as biostimulation. Mitochondrial cytochrome c oxidase is considered as a photoacceptor of low-energy laser. Low-energy He-Ne laser has numberous clinical applications. Our previous studies showed that He-Ne laser irradiation can induce repigmentation in vitiligo vulgaris. However, the exact mechanisms of He-Ne laser irradiation in repigmentation are not elucidated thoroughly. In the past, we have demonstrated the coexistence of both antikertinocyte (anti-KC) and antimelanocyte (anti-MC) IgG antibodies (Abs) in vitiligo patients and explored their potential roles in vitiligo. This current three-year proposal aims to clarify the mechanisms of melanocyte destruction and regeneration in vitiligo lesions using both traditional cell culture and skin equivalent model (organotypic culture). In the first year, we shall focus on the regeneration of MCs and MBs by He-Ne laser with or without the presence of anti-MC IgG antibodies from vitiligo patients, as well as the involved photodynamic mechanisms. Our goal for the second year is to investigate the regeneration of MCs and MBs by He-Ne laser with or without the presence of anti-KC IgG antibodies from vitiligo patients. In the final year of our project, we shall explore the effects of He-Ne laser combine antibody-dependent cellular cytotoxicity (ADCC) on the regeneration of MCs and MBs. Our results will provide more information for the effectiveness of He-Ne laser irradiation in treating vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults and patients with vitiligo

Exclusion Criteria:

* systemic disease

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2005-06; Study Completion 2008-01

PRIMARY OUTCOMES:
foreskin from normal adults

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Su Yu, MD PHD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan